CLINICAL TRIAL: NCT02749630
Title: An Observer-Blinded, Placebo-Controlled, Multiple-Ascending, Dose-Escalation Study to Explore the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Repeat Intravenous Administrations of UTTR1147A in Healthy Volunteers and Patients With Ulcerative Colitis and Crohn's Disease
Brief Title: A Safety Study of Intravenously Administered UTTR1147A in Healthy Volunteers (HVs), Participants With Ulcerative Colitis (UC), and Participants With Crohn's Disease (CD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GA29469; 2015-002512-32 (EudraCT Number)
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Healthy Volunteer (Experimental): Participants will be given escalating doses of UTTR1147A or Placebo intravenously
  Interventions: Drug: Placebo; Drug: UTTR1147A
- Ulcerative Colitis (Experimental): Participants will be given escalating doses of UTTR1147A or Placebo intravenously
  Interventions: Drug: Placebo; Drug: UTTR1147A
- Crohn's Disease (Experimental): Participants will be given escalating doses of UTTR1147A or Placebo intravenously
  Interventions: Drug: Placebo; Drug: UTTR1147A

INTERVENTIONS:
Drug: Placebo — Matching placebo to UTTR1147A administered intravenously
Drug: UTTR1147A — Escalating doses of intravenously administered UTTR1147A
  Other Names: efmarodocokin alfa; RO7021610; RG7880; IL-22Fc

SUMMARY:
This is a randomized, observer-blinded, placebo-controlled study to evaluate safety, tolerability, immunogenicity, and pharmacokinetics of repeat dosing of intravenous (IV) UTTR1147A. The study will consist of a repeat dose escalation in HVs, in participants with UC, and in participants with CD across multiple sites.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* No history of malignancy
* Documentation of age-appropriate cancer screening based on local/country-specific guidelines
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm

For HVs Only:

* Age 18 - 50
* Body mass index (BMI) between 18 and 32 kilograms per square meter (kg/m2), inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), and vital signs, and clinical laboratory evaluations should be within the reference range for the test laboratory unless deemed not clinically significant by the investigator and Sponsor

For Participants with UC or CD:

* Age 18 - 80
* Eligible to receive biologic therapy
* Disease duration of >/= 12 weeks
* Diagnosis of moderate to severe UC or CD

Exclusion Criteria:

General exclusion criteria:

* History of inflammatory skin disorders
* History of any cancer
* History of anaphylaxis, hypersensitivity, or drug allergies
* History of alcoholism or drug addiction
* Positive tests indicating infection for hepatitis C, hepatitis B, or HIV
* Use of a non-biologic investigational drug or participation in an investigational study with a non-biologic drug within 30 days or 5 half-lives of investigational product, whichever is greater, prior to study drug administration
* Use of a biologic investigational therapy or participation in an investigational study involving biologic therapy within 90 days or 5 half-lives, whichever is greater, prior to study drug administration
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion
* Family history of sudden unexplained death or long QT syndrome
* Any acute or chronic condition that would limit the subject's ability to complete and/or participate in this clinical study
* Pregnant or lactating, or intending to become pregnant for duration of study

For HVs Only:

* Known family history of gastrointestinal (GI) and/or colon cancer
* Prior exposure to UTTR1147A

For Participants with UC or CD:

* Significant uncontrolled co-morbidity, such as neurological, cardiac, pulmonary, renal, hepatic, endocrine, or GI disorders
* History of primary sclerosing cholangitis
* Active anti-TNF induced psoriasiform or eczematous lesions
* Moderate to severe anemia
* Presence of an ileostomy or colostomy
* Total proctocolectomy
* Positive screening for latent mycobacterial tuberculosis infection
* Impaired renal function
* Impared hepatic function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Up to Day 134

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of UTTR1147A After the First and Last Dose | Up to Day 134
Minimum (Trough) Serum Concentrations (Ctrough) of UTTR1147A Prior to the Second and Last Dose | Up to Day 134
Total Serum Clearance (CL) of UTTR1147A | Up to Day 134
Volume of Distribution (V) of UTTR1147A | Up to Day 134
Area Under the Concentration vs. Time Curve (AUC) Within a Dose Interval (AUCtau) After the Final Dose of UTTR1147A | Up to Day 134
Elimination Half-Life (t1/2) of UTTR1147A | Up to Day 134
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) in Serum | Up to Day 134

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Charité Research Organisation GmbH, Berlin, Germany
- Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Wagner F, Mansfield JC, Lekkerkerker AN, Wang Y, Keir M, Dash A, Butcher B, Harder B, Orozco LD, Mar JS, Chen H, Rothenberg ME. Dose escalation randomised study of efmarodocokin alfa in healthy volunteers and patients with ulcerative colitis. Gut. 2023 Aug;72(8):1451-1461. doi: 10.1136/gutjnl-2022-328387. Epub 2023 Feb 2. PMID 36732049
- [Derived] Powell N, Pantazi E, Pavlidis P, Tsakmaki A, Li K, Yang F, Parker A, Pin C, Cozzetto D, Minns D, Stolarczyk E, Saveljeva S, Mohamed R, Lavender P, Afzali B, Digby-Bell J, Tjir-Li T, Kaser A, Friedman J, MacDonald TT, Bewick GA, Lord GM. Interleukin-22 orchestrates a pathological endoplasmic reticulum stress response transcriptional programme in colonic epithelial cells. Gut. 2020 Mar;69(3):578-590. doi: 10.1136/gutjnl-2019-318483. Epub 2019 Dec 2. PMID 31792136